CLINICAL TRIAL: NCT04118166
Title: Phase 2 Study of Ipilimumab Plus Nivolumab in Combination With Cryotherapy in Metastatic or Locally Advanced Soft Tissue Sarcoma
Brief Title: Ipilimumab + Nivolumab + Cryotherapy in Metastatic or Locally Advanced Soft Tissue Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kristen Ganjoo (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, Kristen Ganjoo, Associate Professor of Medicine, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-50853; SARCOMA0038 (Other: OnCore)
Record Dates: First submitted 2019-10-02; First posted 2019-10-08 (Actual); Results first posted 2022-10-10 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-11

CONDITIONS: Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Ipilimumab; CTLA-4 Antigen; Cryosurgery; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ipilimumab/nivolumab + cryotherapy (Experimental): 1 mg/kg with nivolumab 3 mg/kg every 3 weeks x 4 doses. (One cycle of treatment is 3 weeks). Cryotherapy (cryoablation) will be performed between investigational agent treatment Cycles 1 and 2
  Interventions: Drug: Ipilimumab; Procedure: Cryoablation; Drug: Nivolumab

INTERVENTIONS:
Drug: Ipilimumab — Ipilimumab 1 mg/kg, injection
  Other Names: Yervoy; BMS-734016; MDX010; MDX-CTLA4
Procedure: Cryoablation — Cryoablation of the tumors occur between investigational agent treatment Cycles 1 and 2, and will be performed according to standard procedures
Drug: Nivolumab — Nivolumab 3 mg/kg, injection
  Other Names: BMS-936558; MDX1106; ONO-4538

SUMMARY:
The purpose of this Phase 2 study is to

1. find out if the study drugs (ipilimumab plus nivolumab) in combination with cryotherapy will help participants with metastatic or locally advanced soft tissue sarcoma;.
2. find out how safe are ipilimumab plus nivolumab given in combination with cryotherapy, and what side effects may be related to treatment.
3. find out how do the study drugs in combination with cryotherapy work in soft tissue sarcoma.

DETAILED DESCRIPTION:
Primary Objectives:

1) Assess whether the rate of clinical benefit is sufficiently high to merit promise for further study

Secondary Objectives:

1. Characterize the 6-month progression-free survival rate
2. Assess whether the treatment yields a reasonably safe and tolerable profile

ELIGIBILITY:
Inclusion Criteria:

* Unresectable or metastatic soft tissue sarcoma
* ≥ 1 prior systemic therapy for sarcoma, including adjuvant systemic therapy
* Age ≥ 18 years
* 4 Life expectancy > 3 months
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Lab values as below:

Absolute neutrophil count (ANC) ≥ 1,000/mm^3 Platelet count ≥ 75,000/mm^3; Creatinine ≤ 1.5 x upper limit of normal (ULN) OR calculated (calc.); creatinine clearance > 45 mL/min using the lean body mass formula only; Total bilirubin ≤ 1.5 x ULN in absence of Gilbert disease (total bilirubin ≤ 3 x ULN with Gilbert); also, if hyperbilirubinemia is clearly attributed to liver metastases total bilirubin ≤ 3 x ULN is permitted AST/ALT ≤ 3 x ULN;Thyroid stimulating hormone (TSH) within normal limits (WNL);supplementation is acceptable to achieve a TSH WNL; in subjects with abnormal TSH if free T4 is normal and subject is clinically euthyroid, subject is eligible

* Any toxic effects of prior therapy (except alopecia) must be resolved to NCI CTCAE, version 5.0, Grade 1 or less
* Ability to understand and the willingness to sign a written informed consent
* Women of childbearing potential (WOCBP) receiving nivolumab must be willing to adhere to contraception for a period of 5 months after the last dose of nivolumab. Men receiving nivolumab and who are sexually active with WOCBP will be instructed and must be willing to adhere to contraception for a period of 7 months after the last dose of nivolumab.

Exclusion Criteria:

* Prior therapy with ipilimumab or nivolumab, or any agent targeting programmed cell death 1 (PD-1), PD-L1 or cytotoxic T-lymphocyte-associated protein 4 (CTLA-4)

History of the following:

* Active known or suspected autoimmune disease
* Known human immunodeficiency virus (HIV) (Subjects with lymphocytes > 350 cluster of differentiation (CD)4+ cells and no detectable viral load are eligible)
* Hepatitis B

Hepatitis B can be defined as:

Hepatitis B surface antigen (HBsAg) > 6 months Serum hepatitis B virus (HBV) deoxyribonucleic acid (DNA) 20,000 IU/mL (105 copies/mL), lower values 2,000 to 20,000 IU/mL (104 to 105 copies/mL) are often seen in hepatitis B-e antigen (HbeAg)-negative chronic hepatitis B Persistent or intermittent elevation in alanine aminotransferase (ALT)/alanine aminotransferase (AST) levels. Liver biopsy showing chronic hepatitis with moderate or severe necroinflammation

* Hepatitis C Hepatitis C antibody (Ab) positive Presence of hepatitis C virus (HCV) ribonucleic acid (RNA) 3.2.2.5 Known active pulmonary disease with hypoxia defined as: Oxygen saturation < 85% on room air or Oxygen saturation < 88% despite supplemental oxygen
* Systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 7 days of registration
* Received any live/attenuated vaccine (eg, varicella, zoster, yellow fever, rotavirus, oral polio and measles, mumps, rubella (MMRI) within 30 days before initiation of treatment on this protocol.
* If female, pregnant or lactating. (Women of childbearing potential are required to have a negative pregnancy test within 24 hours prior to the initial administration of study drug)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Ganjoo, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Medical Center, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ipilimumab/Nivolumab + Cryotherapy
Started | 30
Completed | 29
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ipilimumab/Nivolumab + Cryotherapy
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 8
Age, Continuous [Median (Standard Deviation); unit: years] | 55.0 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 24
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response
Description: Clinical benefit was assessed on the basis of clinical response per the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria:
  * Complete response (CR) = Disappearance of all target lesions; all lymph nodes < 10 mm on the short axis; no new lesions.
  * Partial response (PR) = ≥ 30% decrease in the sum of the longest diameter of target lesions; no new lesions.
  * Stable disease (SD) = Small changes that do not meet any of the above criteria; no new lesions.
  * Progressive disease (PD) = 20% increase in the sum of the longest diameter of target lesions, and/or the appearance of one or more new lesion(s).
  Clinical benefit was defined as CR + PR. The primary outcome is expressed as the total number of participants who receive clinical benefit within 14 weeks, a number without dispersion. Rates of all clinical responses are reported.
Time Frame: 14 weeks
Population: Does not include participants taken off-study, and not evaluated for the outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Ipilimumab/Nivolumab + Cryotherapy
Number analyzed (Participants) | 29
Participants
  Complete Response (CR) | 0
  Partial Response (PR) | 3
  Stable Disease (SD) | 7
  Progressive disease (PD) | 19

2. Secondary Outcome: Related Adverse Events (Toxicity)
Description: Adverse events were assessed per CTCAE version 5. The outcome is those adverse events experienced by participants that were determined to be possibly, probably, or definitely-related to study treatment. Serious adverse events are identified by the term "SAE." Results are presented as the number of related adverse events by preferred term that occurred. The data are numbers without dispersion.
Time Frame: 24 months
Measure: Number; unit: Related adverse events
Groups:
- Number of Occurrences of Related Adverse Events: All adverse events considered to be possibly, probably, or definitely-related to study treatment.
Arm/Group | Number of Occurrences of Related Adverse Events
Number analyzed (Participants) | 30
Related adverse events
  Ringing in the ears (tinnitus) | 1
  Adrenal insufficiency | 1
  Hyperthyroidism (excess levels of thyroxine hormone) | 3
  Hypothyroidism (diminished levels of thyroxine hormone) | 4
  Hypophysitis (inflammation of the pituitary gland) | 1
  Diarrhea | 4
  Diarrhea (intermittent) | 1
  Dry mouth | 2
  Allergic reaction | 1
  Thyroid stimulating hormone (TSH) elevated | 2
  Alanine aminotransferase (ALT) elevated | 1
  Hyponatremia (blood sodium level decreased) | 2
  Neuropathy, peripheral sensory | 1
  Numbness, bilateral hand, intermittent | 1
  Pain, neuropathic | 1
  Cough, all descriptions | 4
  Dyspnea (shortness of breath) | 3
  Hoarse voice | 1
  Pneumonitis (lung inflammation) | 1
  Pneumonitis (lung inflammation) (SAE) | 1
  Rash, all descriptions | 12

3. Secondary Outcome: Immune-related Clinical Response (irRECIST) Rate
Description: The immune-related (ir) clinical response will be assessed per the immune-related Response Evaluation Criteria in Solid Tumors (ir-RECIST) criteria, as follows:
  * Complete response (CR) = Disappearance of all lesions, with any pathological lymph nodes having a reduction in short axis to < 10 mm; no new lesions > 5 × 5 mm in size.
  * Partial response (PR) = ≥ 30% decrease in the sum of the longest diameter of target lesions.
  * Stable disease (SD) = Small changes that do not meet any of the these criteria; no new lesions > 5 × 5 mm in size.
  * Progressive disease (PD) = 20% increase in the sum of the longest diameter of target lesions with the sum of diameters increasing ≥ 5 mm, and/or the appearance of 1+ new lesion(s).
  Note that irRECIST differs from RECIST criteria. The outcome is expressed as the total number of participants who achieve a ir-clinical response (ie, CR + PR) by 16 weeks, a number without dispersion.
Time Frame: 16 weeks
Population: Immune-related Response Evaluation Criteria in Solid Tumors (ir-RECIST) was not assessed/collected for some subjects, and cannot be reported. Reasons that ir-RECIST was not assessed included death, adverse event, and withdrawal/lost-to-follow-up subsequent to PD determination per RECIST at 14 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Ipilimumab/Nivolumab + Cryotherapy
Number analyzed (Participants) | 25
Participants
  Complete response (CR) | 0
  Partial response (PR) | 3
  Stable disease (SD) | 7
  Progressive disease (PD) | 15

4. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival (PFS) is a measure of participants remaining alive without disease progression. The outcome is expressed as the total number of participants remaining alive without disease progression at 6 months after consent, a number without dispersion.
Time Frame: 6 months
Population: Does not include participants taken off-study, and not evaluated for the outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Ipilimumab/Nivolumab + Cryotherapy
Number analyzed (Participants) | 29
Participants | 3

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Ipilimumab/Nivolumab + Cryotherapy
All-Cause Mortality (participants affected / at risk) | 15/30
Serious Adverse Events (participants affected / at risk) | 30/30
Other Adverse Events (participants affected / at risk) | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ipilimumab/Nivolumab + Cryotherapy (N=30)
Anemia (Blood and lymphatic system disorders) | 4 (4)
Cardiac arrest (Cardiac disorders) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1)
Elevated ALT (Investigations) | 2 (3)
Elevated AST (Investigations) | 2 (3)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Other, Disease Progression (death) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 15 (15)
Muscle weakness, right-sided (Nervous system disorders) | 1 (1)
Other, Motor deficit, right side (Nervous system disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Intermittent bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Right apical pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Right pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ipilimumab/Nivolumab + Cryotherapy (N=30)
Anemia (Blood and lymphatic system disorders) | 4 (15)
Other, Deep vein thrombois (DVT) of catheter (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Intermittent heart palpitations (Cardiac disorders) | 2 (2)
Pericarditis (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 2 (2)
Other, Decreased pulse (Cardiac disorders) | 1 (1)
Ringing in the ears (tinnitus) (Ear and labyrinth disorders) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 3 (3)
Hypophysitis (Endocrine disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 4 (4)
Dry eyes (Eye disorders) | 1 (1)
Flashing lights (Eye disorders) | 1 (1)
Intermittent brief blurry vision (Eye disorders) | 1 (1)
Keratitis (Eye disorders) | 1 (1)
L eye redness (Eye disorders) | 1 (1)
L eye pain (Eye disorders) | 1 (1)
L eye burning sensation (Eye disorders) | 1 (1)
L eye blurred vision (Eye disorders) | 1 (1)
R eye blurred vision (Eye disorders) | 1 (1)
Other, Corneal abrasion (Eye disorders) | 1 (1)
Abdominal bloating (Gastrointestinal disorders) | 2 (2)
Intermittent abdominal bloating (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 4 (4)
Increased abdominal pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 3 (4)
Diarrhea (intermittent) (Gastrointestinal disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 5 (6)
Intermittent nausea (Gastrointestinal disorders) | 2 (2)
Intermittent nausea/vomiting (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Other, Decreased appetite (Gastrointestinal disorders) | 3 (3)
Other, Lack of appetite (Gastrointestinal disorders) | 1 (1)
Other, Mucositis (Gastrointestinal disorders) | 1 (1)
Chest Pain (General disorders) | 1 (1)
Fatigue (General disorders) | 9 (9)
Fever (General disorders) | 4 (4)
Intermittent fever (General disorders) | 1 (1)
Low grade fever (General disorders) | 1 (1)
Flu-like symptoms (General disorders) | 1 (1)
Intermittent chest pain to R sternal border exacerbated with deep inhalation (General disorders) | 1 (1)
Intermittent fatigue (General disorders) | 1 (1)
Intermittent chills followed by hot flashes (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1)
Gum infection (Infections and infestations) | 1 (1)
UTI (Infections and infestations) | 1 (1)
Other, Infectious diarrhea (Infections and infestations) | 1 (1)
Other, Presumed pneumonia (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Elevated TSH (Investigations) | 1 (1)
TSH increased (Investigations) | 1 (1)
Decreased WBC count (Investigations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1)
Elevated ALT (Investigations) | 1 (1)
Weight loss (Investigations) | 4 (4)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthralgias (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle and joint aches (Musculoskeletal and connective tissue disorders) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Lower back throbbing pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Right neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Right shoulder pain (Pain in extremity) (Musculoskeletal and connective tissue disorders) | 1 (1)
Other, Gluteal pain and swelling (Musculoskeletal and connective tissue disorders) | 1 (1)
Other, Arm pain left (Musculoskeletal and connective tissue disorders) | 1 (1)
Other, Muscle aches and fatigue associated with COVID vaccine (Musculoskeletal and connective tissue disorders) | 1 (1)
Other, Right thigh pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Other, Soreness to right lateral ribs (Musculoskeletal and connective tissue disorders) | 1 (1)
Other, Soreness at site of recent cryoablation (R lung) (Musculoskeletal and connective tissue disorders) | 1 (1)
Other, Soreness right chest wall (Musculoskeletal and connective tissue disorders) | 1 (1)
Other, Soreness to left side at site of recent cryoablation (Musculoskeletal and connective tissue disorders) | 1 (1)
Other, Soreness, right shoulder (Musculoskeletal and connective tissue disorders) | 1 (1)
Other, Pain to right chest wall at recent site of cryo (Musculoskeletal and connective tissue disorders) | 2 (2)
Other, Pelvic bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Other, Intermittent peripheral edema (Musculoskeletal and connective tissue disorders) | 1 (1)
Other, Weakness to left shoulder (Musculoskeletal and connective tissue disorders) | 1 (1)
Worsening left leg weakness (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Muscle weakness, left-sided (Nervous system disorders) | 1 (1)
Muscle weakness, right-sided (Nervous system disorders) | 1 (1)
Neuropathy under R axilla (Nervous system disorders) | 1 (1)
Other, Intermittent bilateral hand numbness (Nervous system disorders) | 1 (1)
Other, Motor deficit, left side (Nervous system disorders) | 1 (1)
Other, Motor deficit, right side (Nervous system disorders) | 1 (1)
Other, Neuropathic pain (Nervous system disorders) | 1 (1)
Other, Occasional twitching sensation to anterior chest wall (Nervous system disorders) | 1 (1)
Other, Intermittent left sciatic pain (Nervous system disorders) | 1 (1)
Worsening anxiety (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Intermittent hematuria (Renal and urinary disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Blood tinge sputum (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (8)
Intermittent cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Intermittent cough w/chest tightness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Intermittent cough with Blood tinge sputum (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dry cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Worsening cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Shortness of breath with exertion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hoarse voice (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Right pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Right apical pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Tension pneumothorax (requiring ICU stay) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper respiratory infection (COVID-19) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Intermittent wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Other, Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Facial rash (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 4 (4)
Maculo-papular rash (Skin and subcutaneous tissue disorders) | 1 (1)
Maculo-papular rash to bilateral arms (Skin and subcutaneous tissue disorders) | 1 (1)
Post-inflammatory hyperpigmentation on left breast (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 5 (5)
Tinea (Skin and subcutaneous tissue disorders) | 1 (1)
Other, Burned hand (Skin and subcutaneous tissue disorders) | 1 (1)
Other, Hair thinning (Skin and subcutaneous tissue disorders) | 1 (1)
Other, Leg ulcer left (Skin and subcutaneous tissue disorders) | 1 (1)
Other, Molluscum contagiousum on left arm (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-26): https://cdn.clinicaltrials.gov/large-docs/66/NCT04118166/Prot_SAP_000.pdf